CLINICAL TRIAL: NCT05203146
Title: Assessing the Impact of a Mobile Device App to Improve Emergency Care Efficiency and Remote Collaborative and Synchronous Communication in a Pediatric Emergency Department: a Pilot Randomized Controlled Trial
Brief Title: PIMPmyHospital: a Mobile App to Improve Emergency Care Efficiency and Communication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pediatric Clinical Research Platform (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Johan Siebert, MD, MD, Deputy Head, Pediatric Clinical Research Platform
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PIMPmyHospital
Record Dates: First submitted 2022-01-07; First posted 2022-01-24 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Pediatric Emergency Medicine; Communication
Keywords: Information technologies; Mobile Applications; Laboratory Result Delivery; Information Storage and Retrieval; Hospital Communication Systems; Communication; Pediatric Emergency Medicine; Emergency Department
MeSH Terms: conditions — Communication; Emergencies

STUDY DESIGN:
Intervention Model Description: A prospective, single center, randomized, controlled trial
Who Masked: Participant
Masking Description: Blinding to the outcomes will be maintained during recruitment to minimize preparation bias. Allocation concealment will be ensured with an allocation software (www.sealedenvelope.com) and will not be released until the participants start the scenario. A post-scenario review will be done without blinding by two study investigators, but undertaken independently with each blinded to the other's reviews. In the case of disagreement, a third independent evaluator will help reach a consensus. The data analyst will not be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (PIMPmyHospital) (Experimental): Participants that will use the mobile heath PIMPmyHospital tool during the semi-simulation-based scenario.
  Interventions: Device: PIMPmyHospital (mobile health tool)
- Arm B (Conventional methods) (Active Comparator): Participants that will use conventional methods (i.e., without mobile app support) during the semi-simulation-based scenario.
  Interventions: Other: Conventional method

INTERVENTIONS:
Device: PIMPmyHospital (mobile health tool) — Each participant will first be asked to retrieve a factious patient's laboratory results on the app when randomly made available, and then reach a colleague (role played by a study investigator) when asked to do so by a text message on the app.
  Arms: Arm A (PIMPmyHospital)
Other: Conventional method — Each participant will first be asked to retrieve a factious patient's laboratory results from the emergency department's computerized patient data system when randomly made available, and then contact a colleague (role played by a study investigator) when asked to do so (request made by a second study investigator).
  Arms: Arm B (Conventional methods)

SUMMARY:
This pilot study is a prospective, single-center, randomized, controlled trial in a tertiary pediatric emergency department with two parallel groups of voluntary post-graduate year 1 to 5 pediatric residents and registered pediatric emergency nurses. The impact of an mHealth support tool will be compared to conventional methods on the retrieval of laboratory data from the patient's electronic record, and on team collaboration in a semi-simulated emergency department environment. Ten participants are randomized (1:1). The primary endpoint is the time from the availability of new laboratory results for a given patient to their consideration by participants, measured in minutes using a stopwatch.

DETAILED DESCRIPTION:
Emergency care is very complex in that it requires patient-centered care in a coordinated manner among multiple providers in a highly distractible, unpredictable, multi-tasking, and stressful environment. Due to the inherent characteristics of specimen processing and laboratory instruments, the turnaround time from laboratory test ordering to availability of results can be long. As a result, caregivers must continue their multiple tasks while waiting for these results and, in the absence of reminder alerts, they must remember to check their availability. This can lead to oversights or delays in their consideration. Lack of follow-up of abnormal laboratory results can lead to missed information that could impact patient care and safety. Moreover, sharing information efficiently between providers in this environment is difficult. Caregivers are often far away from each other, busy with their tasks, without the ability to quickly communicate face-to-face with their colleagues to exchange important information regarding their patients.

Connecting emergency service providers to each other through a digital communication channel could improve the efficiency of synchronous information sharing and emergency care, as well as instant retrieval of laboratory results at the point of care. To this end, the investigators have developed a mobile application (app) dedicated to emergency department caregivers, PIMPmyHospital (Patients In My Pocket in my Hospital [PubMed Identifier number 34734879]). This app aims to provide relevant information in real time about the patients emergency departments' caregivers are caring for, including laboratory results, as well as a chat and secure messaging platform to virtually connect physicians and nurses caring for the same patients.

This clinical trial is a pilot, prospective, single-center, randomized, controlled trial in a tertiary pediatric emergency department (>33,000 consultations/year) with two parallel groups of voluntary PGY 1 to 5 pediatric residents and registered pediatric emergency nurses. It aims to assess the impact of the app in a real pediatric emergency department environment through standardized, semi-simulated scenarios. Ten participants (5 residents and 5 nurses) are randomized 1:1.

During their actual clinical tasks, each participant is asked to take note of laboratory results about a fictional patient that randomly occur once during the course of the scripted scenario, using either the app (study arm A) or conventional methods (study arm B), and secondly, to then respond to requests from a remote colleague to go to a specific location in the emergency room to assist with a technical procedure (the request being relayed either by the app or one of the study investigators depending on the study arm allocation).

The primary endpoint is the time from the availability of new laboratory results to their consideration by participants, measured in minutes using a stopwatch.

The secondary endpoint is the time from when the participant is informed that a colleague requires his or her assistance to perform a technical procedure to when the participant reaches that colleague, measured in minutes using a stopwatch.

Data collection is carried out by two study investigators. Deidentified data are safely stored in duplicate on papers and secured hard-disk drives in a locked room at the Geneva Children's Hospital, Switzerland. This study offers the major advantage to observe a unique period per participant during their regular shift. Therefore, neither follow-up nor retention plans is necessary. The REDCap database (REDCap, Vanderbilt University, Nashville, Tennessee, USA) will be used for data collection. Study data will be de-identified and a master linking log (code key) with identifiers (ie, participant identification list on paper format) will be kept and stored separately from the data by the study investigators in a secured cabinet in a locked room at Geneva Children's Hospital, Switzerland, under the responsibility of the principal investigator.

This clinical trial will assess the impact of a collaborative mHealth tool to increase timely medical information retrieval at the point of care and team communication in an emergency department. The results of this pilot study will be used to set up a larger randomized controlled trial. As research in this area is scarce, the results generated from this study could be of importance to improve in-hospital pediatric emergency care practice and communication in an era of communication technologies.

ELIGIBILITY:
Inclusion Criteria:

* Any postgraduate residents pursuing a <6 years residency in pediatrics.
* To be registered nurses from the pediatric emergency department.
* To have previously completed a standardized 5-min introductory course on the use of the PIMPmyHospital tool dispensed by the study investigators.
* Participation agreement.

Exclusion Criteria:

* To have not undergone the standardized 5-min introductory course on the use of the PIMPmyHospital tool dispensed by the study investigators.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2021-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johan N Siebert, MD, Principal Investigator — Geneva Children's Hospital, Geneva University Hospitals, Geneva, Switzerland
Locations (1):
- Geneva Children's Hospital, Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data will be deidentified and the study investigators will house the data locally on paper files and secure hard disk drives at the Geneva Children's Hospital. The datasets used or analyzed during the current trial will be available from the corresponding author upon reasonable request, recognizing that these data will only provide results for the current pilot trial and not for future randomized controlled trials that would follow. Only deidentified/anonymized data will be shared.
Supporting Information: Study Protocol
Time Frame: Available from 6 month to 5 years after trial publication.
Access Criteria: * Data will be made available from the corresponding author upon approval of a proposal and with a signed data access agreement.
  * Deidentified participant data will be made available to qualified external researchers whose proposed use of the data has been approved by their Institutional Review Board.
  * Data will be made available for a specified research purpose.
  * The request proposal must include a statistician.

REFERENCES:
- [Result] Ehrler F, Tuor C, Rey R, Siebert JN. A Mobile App to Improve Patient Management in Emergency Departments: Caregiver Needs Analysis, Design and Early Technology Acceptance Assessment. Stud Health Technol Inform. 2021 Oct 27;285:233-238. doi: 10.3233/SHTI210605. PMID 34734879
- [Result] Ehrler F, Tuor C, Trompier R, Berger A, Ramusi M, Rey R, Siebert JN. Effectiveness of a Mobile App in Reducing Therapeutic Turnaround Time and Facilitating Communication between Caregivers in a Pediatric Emergency Department: A Randomized Controlled Pilot Trial. J Pers Med. 2022 Mar 9;12(3):428. doi: 10.3390/jpm12030428. PMID 35330427

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (PIMPmyHospital) | Arm B (Conventional Methods)
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A (PIMPmyHospital): Participants that will use the mHeath PIMPmyHospital tool during the semi-simulation-based scenario.
  PIMPmyHospital (mHealth tool): Each participant will first be asked to retrieve a factious patient's laboratory results on the app when randomly made available, and then reach a colleague (role played by a study investigator) when asked to do so by a text message on the app.
- Total: Total of all reporting groups
Arm/Group | Arm A (PIMPmyHospital) | Arm B (Conventional Methods) | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (8.5) | 30.8 (3.7) | 32.5 (6.4)
Age, Customized [Count of Participants; unit: Participants] — Age in years, n (%)
  Participants
    <30 | 1 | 2 | 3
    30-39 | 3 | 3 | 6
    >=40 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Work experience since certification [Mean (Standard Deviation); unit: years] | 10.8 (9.1) | 5.8 (3.4) | 8.5 (7.1)
Work experience since certification [Count of Participants; unit: Participants]
  <5 | 1 | 2 | 3
  5-9 | 2 | 2 | 4
  >=9 | 2 | 1 | 3
Work experience in the Pediatric Emergency Department [Mean (Standard Deviation); unit: months] | 69.3 (72.7) | 36.6 (26.6) | 53.0 (54.4)
Work experience in the Pediatric Emergency Department [Count of Participants; unit: Participants]
  <12 | 1 | 1 | 2
  12-24 | 1 | 1 | 2
  >=24 | 3 | 3 | 6
Satisfaction with current timelines from laboratory report to review, [Mean (Standard Deviation); unit: units on a scale] — on a 10-point Likert scale (0 = not at all satisfied, 10 = extremely satisfied)
  units on a scale | 4.4 (1.1) | 5.0 (2.2) | 4.7 (2.2)
Satisfaction with current situation to find a peer [Mean (Standard Deviation); unit: units on a scale] — on a 10-point Likert scale (0 = not at all satisfied, 10 = extremely satisfied)
  units on a scale | 3.6 (0.5) | 2.2 (1.8) | 2.9 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Time to Laboratory Results
Description: Time elapsed between the availability of new laboratory results on either the mobile app or the pediatric emergency department's computerized patient data system and their consideration by the participant on the allocated medium (i.e., the mobile app or computerized patient data system), measured using a stopwatch.
Time Frame: minutes (upper bound arbitrarily set at 2 hours)
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Arm A (PIMPmyHospital) | Arm B (Conventional Methods)
Number analyzed (Participants) | 5 | 5
Minutes | 1 [0.0 to 5.0] | 23 [10.5 to 49.0]

2. Secondary Outcome: Time to Reach Colleagues
Description: The elapsed time (in minutes) from the moment the participant was informed by the mobile app or a statement given by a study investigator (conventional method) that a nurse required assistance to perform a technical procedure up to the point in time when the participant reached that nurse.
Time Frame: minutes (upper bound arbitrarily set at 2 hours)
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Arm A (PIMPmyHospital) | Arm B (Conventional Methods)
Number analyzed (Participants) | 5 | 5
Minutes | 1 [0.0 to 3.5] | 24 [2.5 to 43.0]

ADVERSE EVENTS:
Time Frame: 0
Description: As it is a simulation-based study, deaths and adverse events were not collected
Arm/Group | Arm A (PIMPmyHospital) | Arm B (Conventional Methods)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT05203146/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT05203146/SAP_001.pdf